CLINICAL TRIAL: NCT06285864
Title: Sense to Act: Pilot Randomized-controlled Trial of an Interoceptive Sensibility Intervention for Musculoskeletal Pain
Brief Title: Sense to Act: An Interoceptive Sensibility Intervention for Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iscte-University Institute of Lisbon (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other); University of Évora (Other)
Responsible Party: Principal Investigator, Ines Oliveira, MSc, Iscte-University Institute of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 122/2023
Record Dates: First submitted 2024-02-01; First posted 2024-02-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-04

CONDITIONS: Musculoskeletal Pain; Chronic Pain
Keywords: interoception; musculoskeletal pain; feasibility
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be unaware of their assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interoception-based intervention (Experimental): The interoception-based intervention group will receive the intervention, which consists of 8 weekly sessions, of 1h30 hour, in groups (4-8 participants in each group).
  Interventions: Behavioral: Interoception-based intervention
- Waiting list (No Intervention): The waiting list group will maintain their treatments as usual and receive the interoception-based intervention, at the end of the study.

INTERVENTIONS:
Behavioral: Interoception-based intervention — Intervention will include body awareness, sensorial, and relaxation exercises, plus homework.
  Arms: Interoception-based intervention

SUMMARY:
The ability to be connected and act according to bodily information is fundamental in chronic pain adjustment. This study aims to test the feasibility of an intervention designed to improve interoceptive sensibility, i.e., the ability to sense, interpret, and regulate bodily sensations in chronic musculoskeletal pain patients.

DETAILED DESCRIPTION:
Background: Interoceptive sensibility (IS), the self-reported experience of internal states, involves individuals' capacity to sense, interpret, integrate, and regulate their own bodily information. Disruptions in interoceptive processes are often associated with various health conditions, including mental illness and chronic pain (CP). Individuals with chronic musculoskeletal pain present disruptions in IS associated with worse pain adjustment.

While there is a growing body of research testing interoceptive-based interventions on both healthy and clinical samples, interventions specifically tailored for individuals with CP are limited. Furthermore, despite evidence that interventions such as mindfulness or meditation improve IS in incividuals with CP, the mechanisms contributing to enhanced pain-related outcomes remain unknown. Additionally, in Portugal, there is a lack of cost-effective interventions for CP in both public health services and the community.

This study aims to address these gaps by evaluating the feasibility of a program designed for a community setting. The program is specifically developed to enhance IS, potentially improving pain adjustment in individuals with chronic musculoskeletal pain - one of the most prevalent and burdensome types of pain globally. The study compares a group receiving an interoception-based intervention, intending to improve IS, against a control group on a waiting list, examining the intervention's acceptability, feasibility, appropriateness, and estimated treatment effects.

Method: The recruitment process will be conducted through the study website, providing information about the research team, study objectives, and general details about the intervention structure and session schedules. Potential participants must register on the website to enroll in the study. Measurements will be collected anonymously and online (via Qualtrics) using self-report questionnaires at four points in time: before (T0), in the middle (T1), at the end (T2), and one month after the intervention (T3). Additionally, participants in the intervention group will complete an anonymous evaluation checklist after each session and a final evaluation checklist assessing the study's acceptability, appropriateness, and feasibility. Block-stratified randomization of participants for each group (intervention/control), based on sex and geographical area (Lisbon/Évora), will be conducted using randomization software.

The intervention includes four stages addressing different IS skills with 8 weekly sessions (4-6 participants), each lasting 1.5 hours. These sessions will be delivered by two trained psychomotor therapists with clinical experience, supplemented by daily home exercises. To ensure fidelity of the procedures during sessions, recordings will be made for later review (therapists cross-confirm each other's sessions).

Discussion: It is expected that, with or without protocol modifications: 1) The protocol components are suitable to conduct a larger study; 2) the program has good acceptability, appropriateness, feasibility, and participant adherence.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals (over 18 years old)
* experiencing chronic musculoskeletal pain (≥ 3 months)
* able to understand and speak portuguese

Exclusion Criteria:

* neurodegenerative diseases
* cancer pain
* recent fractures, or surgeries (< 3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-02-11 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility - Sessions' acceptability | Up to 24 hours after each intervention session.
  Session evaluation checklist - 7 questions answered on a 5-point scale ranging from 1 (totally disagree) to 5 (completely agree), plus 1 open question asking for improvement suggestions.
Feasibility - Program acceptability, appropriateness, and feasibility | Up to 72 hours after the end of the intervention (T2)
  Program evaluation checklist: 21 questions answered on a 5-point scale ranging from 1 (totally disagree) to 5 (completely agree) plus 3 open questions.
Feasibility - Recruitment, retention, and attendance rates | Up to 12 weeks after the end of the intervention
  Number of participants recruited, number of participants included in the study (among those who are eligible), and average number of sessions attended in intervention by participants.
Feasibility - safety/unexpected events | Up to 12 weeks after the end of the intervention
  Number and type of unexpected events reported by the participants during their participation in the intervention.
Feasibility - Treatment Fidelity Check | Up to 12 weeks after the end of the intervention.
  Sessions will be audio-recorded and an independent therapist will confirm if planned procedures were done.

SECONDARY OUTCOMES:
Interoceptive sensibility | Within the 72-hour period before the first session (T0); up to 72 hours after the fourth session (T1), up to 72 hours after the last (eighth) session (T2), and one month after the last session (T3).
  Multidimensional Assessment of Interoceptive Awareness assesses IS skills, such as identifying bodily sensations, body-mind relationships, and body trust, through 32 items rated on a 6-point Likert scale. Higher scores expresses higher IS levels.
Psychological flexibility | Within the 72-hour period before the first session (T0); up to 72 hours after the fourth session (T1), up to 72 hours after the last (eighth) session (T2), and one month after the last session (T3).
  The Portuguese Comprehensive Assessment of Acceptance and Commitment Therapy Processes is an 18-item scale that measures psychological flexibility (openness to experience, behavioral awareness, valued action) on a 7-point rating scale. Higher scores indicate greater psychological flexibility.
Emotion regulation | Within the 72-hour period before the first session (T0); up to 72 hours after the fourth session (T1), up to 72 hours after the last (eighth) session (T2), and one month after the last session (T3).
  Difficulties in Emotion Regulation Scale - Short Form assesses difficulties in emotion regulation (e.g., nonacceptance of emotional responses, difficulty engaging in goal-directed behavior or in impulse control, lack of emotional awareness), through 18 items. Higher scores correspond to more difficulty in emotion regulation.
Pain-related self-efficacy | Within the 72-hour period before the first session (T0); up to 72 hours after the fourth session (T1), up to 72 hours after the last (eighth) session (T2), and one month after the last session (T3).
  The Pain Self-Efficacy Questionnaire assesses the individuals' confidence level in reaching activities or goals, despite pain with 10 items rated on a 7-point scale. Higher scores represent higher self-efficacy levels.
Pain catastrophizing | Within the 72-hour period before the first session (T0); up to 72 hours after the fourth session (T1), up to 72 hours after the last (eighth) session (T2), and one month after the last session (T3).
  Pain Catastrophizing Scale measures pain-related catastrophic thinking through 13 items rated on a 5-point scale.Higher levels express higher levels of pain catastrophizing.
Activity patterns | Within the 72-hour period before the first session (T0); up to 72 hours after the fourth session (T1), up to 72 hours after the last (eighth) session (T2), and one month after the last session (T3).
  Activity Patterns Scale measures activity patterns through 24 questions responded to on a 5-point scale (avoidance, persistence, and pacing related patterns). Higher levels represent more use of the respective pattern.
Affective distress (depression and anxiety) | Within the 72-hour period before the first session (T0); up to 72 hours after the fourth session (T1), up to 72 hours after the last (eighth) session (T2), and one month after the last session (T3).
  Depression Anxiety Stress Scales evaluate depression/anxiety/stress levels experienced during the previous week, through 21 items rated on a 4-point scale. Higher levels represent higher depression and anxiety levels.
Pain severity | Within the 72-hour period before the first session (T0); up to 72 hours after the fourth session (T1), up to 72 hours after the last (eighth) session (T2), and one month after the last session (T3).
  Brief Pain Inventory assesses pain-related disability (e.g., general activities, walking, work, mood) through 7 items rated on 11-point numerical scales; Graded Chronic Pain Scale-Revised (Von Korff et al., 2020) identify chronic pain individuals, grading their pain severity, through 6 items.
Physical function and Vitality | Within the 72-hour period before the first session (T0); up to 72 hours after the fourth session (T1), up to 72 hours after the last (eighth) session (T2), and one month after the last session (T3).
  Medical Outcomes Study-36 - Short Form 36v2 assesses functional limitations in daily physical activities, and vitality, through 10 and 4 items, rated on 4 and 5-point scales, respectively. Higher scores correspond to higher physical function and vitality.

CONTACTS AND LOCATIONS:
Overall Officials: Inês Oliveira, MSc, Principal Investigator — Iscte-University Institute of Lisbon; Sónia Bernardes, PhD, Study Chair — Iscte-University Institute of Lisbon; Margarida Garrido, PhD, Study Chair — Iscte-University Institute of Lisbon
Locations (2):
- Portugal (2):
  - Iscte - University Institute of Lisbon, Lisbon, Lisbon District
  - University of Évora, Evora, Évora District

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication will be made available upon request (De-identified).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study publication.
Access Criteria: Researchers interested in accessing the IPD for further analysis or collaboration should submit a formal request to the authors. Requests will be evaluated based on ethical considerations, data access criteria, and adherence to data use agreements.

REFERENCES:
- [Background] Ferreira PL. [Development of the Portuguese version of MOS SF-36. Part I. Cultural and linguistic adaptation]. Acta Med Port. 2000 Jan-Apr;13(1-2):55-66. Portuguese. PMID 11059056
- [Background] Ferreira PL. [Development of the Portuguese version of MOS SF-36. Part II --Validation tests]. Acta Med Port. 2000 May-Jun;13(3):119-27. Portuguese. PMID 11026151
- [Background] Sullivan, M. J. L., Bishop, S. R., & Pivik, J. (1995). The Pain Catastrophizing Scale: Development and validation. Psychological Assessment, 7(4), 524-532. https://doi.org/10.1037/1040-3590.7.4.524
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Psychometric properties of the portuguese version of the Pain Self-Efficacy Questionnaire. Acta Reumatol Port. 2011 Jul-Sep;36(3):260-7. PMID 22113601
- [Background] Kaufman EA, Xia M, Fosco G, Yaptangco M, Skidmore CR, Crowell SE. The Difficulties in Emotion Regulation Scale Short Form (DERS-SF): Validation and replication in adolescent and adult samples. Journal of Psychopathology and Behavioral Assessment. 2016;38(3):443-455. doi: 10.1007/s10862-015-9529-3.
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Azevedo LF, Altamiro CP, Cláudia D, Luís A, Laurinda L, José R, Teresa P, Sílvia VS, Rosário A, Carlos JC, Maria CC, Duarte C, José C, Georgina C, Beatriz CL, Maria CL, Beatriz S, José CL. Tradução, adaptação cultural e estudo multicêntrico de validação de instrumentos para rastreio e avaliação do impacto da dor crónica. Dor 2007;15:6-56.
- [Background] Cleeland CS. Measurement of pain by subjective report. Advances in pain research and therapy: issues in pain measurement. Vol. 12. New York, NY: Raven Press, 1989. p. 391-403.
- [Background] Pais-Ribeiro J, Honrado A, Leal I. Contribuição para o estudo da adaptação portuguesa das Escalas de Ansiedade, Depressão e Stress (EADS) de 21 itens de Lovibond e Lovibond. Psicol Saúde Doenc¸ as 2004; 5:229-39.
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Von Korff M, DeBar LL, Krebs EE, Kerns RD, Deyo RA, Keefe FJ. Graded chronic pain scale revised: mild, bothersome, and high-impact chronic pain. Pain. 2020 Mar;161(3):651-661. doi: 10.1097/j.pain.0000000000001758. PMID 31764390
- [Background] Esteve R, Ramirez-Maestre C, Peters ML, Serrano-Ibanez ER, Ruiz-Parraga GT, Lopez-Martinez AE. Development and Initial Validation of the Activity Patterns Scale in Patients With Chronic Pain. J Pain. 2016 Apr;17(4):451-61. doi: 10.1016/j.jpain.2015.12.009. Epub 2015 Dec 23. PMID 26724275
- [Background] Mehling WE, Price C, Daubenmier JJ, Acree M, Bartmess E, Stewart A. The Multidimensional Assessment of Interoceptive Awareness (MAIA). PLoS One. 2012;7(11):e48230. doi: 10.1371/journal.pone.0048230. Epub 2012 Nov 1. PMID 23133619
- [Background] Machorrinho J, Veiga G, Fernandes J, Mehling W, Marmeleira J. Multidimensional Assessment of Interoceptive Awareness: Psychometric Properties of the Portuguese Version. Percept Mot Skills. 2019 Feb;126(1):87-105. doi: 10.1177/0031512518813231. Epub 2018 Nov 19. PMID 30451581
- [Background] Cimmino MA, Ferrone C, Cutolo M. Epidemiology of chronic musculoskeletal pain. Best Pract Res Clin Rheumatol. 2011 Apr;25(2):173-83. doi: 10.1016/j.berh.2010.01.012. PMID 22094194
- [Background] Oliveira I, Garrido MV, Bernardes SF. On the body-mind nexus in chronic musculoskeletal pain: A scoping review. Eur J Pain. 2022 Jul;26(6):1186-1202. doi: 10.1002/ejp.1944. Epub 2022 Apr 4. PMID 35315163
- [Background] Bonaz B, Lane RD, Oshinsky ML, Kenny PJ, Sinha R, Mayer EA, Critchley HD. Diseases, Disorders, and Comorbidities of Interoception. Trends Neurosci. 2021 Jan;44(1):39-51. doi: 10.1016/j.tins.2020.09.009. PMID 33378656
- [Background] Khalsa SS, Adolphs R, Cameron OG, Critchley HD, Davenport PW, Feinstein JS, Feusner JD, Garfinkel SN, Lane RD, Mehling WE, Meuret AE, Nemeroff CB, Oppenheimer S, Petzschner FH, Pollatos O, Rhudy JL, Schramm LP, Simmons WK, Stein MB, Stephan KE, Van den Bergh O, Van Diest I, von Leupoldt A, Paulus MP; Interoception Summit 2016 participants. Interoception and Mental Health: A Roadmap. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jun;3(6):501-513. doi: 10.1016/j.bpsc.2017.12.004. Epub 2017 Dec 28. PMID 29884281
- [Background] Hilton L, Hempel S, Ewing BA, Apaydin E, Xenakis L, Newberry S, Colaiaco B, Maher AR, Shanman RM, Sorbero ME, Maglione MA. Mindfulness Meditation for Chronic Pain: Systematic Review and Meta-analysis. Ann Behav Med. 2017 Apr;51(2):199-213. doi: 10.1007/s12160-016-9844-2. PMID 27658913
- [Background] Chen WG, Schloesser D, Arensdorf AM, Simmons JM, Cui C, Valentino R, Gnadt JW, Nielsen L, Hillaire-Clarke CS, Spruance V, Horowitz TS, Vallejo YF, Langevin HM. The Emerging Science of Interoception: Sensing, Integrating, Interpreting, and Regulating Signals within the Self. Trends Neurosci. 2021 Jan;44(1):3-16. doi: 10.1016/j.tins.2020.10.007. PMID 33378655
- [Background] Moreira, H., Gouveia, M. J., & Canavarro, M. C. (2022). A bifactor analysis of the Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) in a sample of adolescents and adults. Current Psychology, 41(2), 757-782. https://doi.org/10.1007/s12144-019-00602-5
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Trindade, I. A., Ferreira, N. B., Mendes, A. L., Ferreira, C., Dawson, D., & Golijani-Moghaddam, N. (2021). Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT): Measure refinement and study of measurement invariance across Portuguese and UK samples. Journal of Contextual Behavioral Science, 21, 30-36. https://doi.org/10.1016/j.jcbs.2021.05.002
- [Background] Francis, A. W., Dawson, D. L., & Golijani-Moghaddam, N. (2016). The development and validation of the Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT). Journal of Contextual Behavioral Science, 5(3), 134-145. https://doi.org/10.1016/j.jcbs.2016.05.003
- [Background] Trindade, I. A., Vagos, P., Moreira, H., Fernandes, D. V., & Tyndall, I. (2022). Further validation of the 18-item Portuguese CompACT scale using a multi-sample design: Confirmatory factor analysis and correlates of psychological flexibility. Journal of Contextual Behavioral Science, 25, 1-9. https://doi.org/10.1016/j.jcbs.2022.06.003